CLINICAL TRIAL: NCT06081595
Title: Fluzoparib Combined With Apatinib for Maintenance Treatment in Platinum-Sensitive Relapsed Ovarian Carcinoma: A Phase II Single-arm, Open Label, Multicenter Trial
Brief Title: Fluzoparib Combined With Apatinib in Relapsed Ovarian Carcinoma Maintenance Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jin Li (Other)
Responsible Party: Sponsor-Investigator, Jin Li, MD, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-OC-II-011
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Relapsed Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — fluzoparib; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluzoparib+Apatinib combination (Experimental)
  Interventions: Drug: Fluzoparib; Drug: Apatinib

INTERVENTIONS:
Drug: Fluzoparib — Fluzoparib 100mg bid
Drug: Apatinib — Apatinib 375mg qd

SUMMARY:
This study is a Phase II single-arm, open label, multicenter study to access the effects and tolerability of fluzoparib combined with apatinib for maintenance treatment in platinum-sensitive relapsed ovarian carcinoma .

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily joined the study and signed the informed consent.
* Age 18-75 years old.
* Participant has histologically confirmed diagnosis of high-grade predominantly serous ovarian cancer, fallopian tube cancer, primary peritoneal cancer; Or moderately or poorly differentiated ovarian endometrioid adenocarcinoma.
* Previously, after undergoing 2-3 lines of platinum containing chemotherapy, CR or PR was achieved, and the time from the penultimate platinum containing chemotherapy to PD was ≥ 6 months.
* Patients who have received previous treatment with bevacizumab are acceptable.
* Allow previous treatment with PARP inhibitors other than Fluzoparib.
* ECOG score: 0-1.
* Participant has adequate organ function as defined in the following contents (Any blood component or cell growth factor within 14 days prior to randomization is not permitted) Absolute neutrophil count (ANC) ≥1.5×109/L Platelets ≥100×109/L Hemoglobin ≥10g/dL Serum albumin ≥3g/dL Total bilirubin ≤1.5 ×ULN AST (SGOT) and ALT (SGPT) ≤3 × ULN Serum creatinine ≤1.5 × ULN
* Patients with potential fertility need to use a medically approved contraceptive (such as an intrauterine device, birth control pill or condom) during he study treatment period and within 2 months after the last administration of apatinib or 6 months after the last administration of fluzopril, whichever is longer; Serum HCG or urine HCG must be negative within 72 hours prior to study enrollment; must be a non-lactation period.

Exclusion Criteria:

* Previous (within 5 years) or concurrent with other uncured malignant tumors, except for cured skin basal cell carcinoma, thyroid cancer, cervical carcinoma in situ and breast cancer with no recurrence >3 years after radical surgery.
* The subject has untreated central nervous system metastasis.
* Inability to swallow pills normally, or gastrointestinal dysfunction, which may affect drug absorption according to the researchers.
* Recent (within 3 months) occurrence of intestinal obstruction.
* Patients with clinical symptoms of cancerous ascites and pleural effusion, who need puncture or drainage, or who have received ascites and pleural effusion drainage within 2 months before the first trial medication.
* Patients with poorly controlled cardiac clinical symptoms or diseases, such as: (1) NYHA2 or higher heart failure, (2) unstable angina pectoris, (3) myocardial infarction within 1 year, (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention, (5) QTc>470ms.
* Those with abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds), who have a bleeding tendency or are receiving thrombolytic or anticoagulant therapy, are allowed to receive low-dose low-molecular weight heparin or oral aspirin prophylactic anticoagulant therapy during the trial.
* The subject has an active infection or unexplained fever >38.5 degrees during the screening period and before the first dose;
* Subjects with congenital or acquired immune deficiency (such as HIV infection), or active hepatitis (hepatitis B reference: HBsAg positive and HBV DNA≥500 IU/ml; Hepatitis C reference: HCV antibody positive and HCV copy number > upper limit of normal).
* Those who had previously received radiotherapy, chemotherapy, endocrine therapy, or molecular targeted therapy and were enrolled less than 4 weeks after the completion of treatment (last dose); Adverse events (except alopecia) caused by previous treatment did not recover to ≤1 degree (CTCAE 5.0).
* Patients who have used other drugs in clinical trial studies within the previous 4 weeks.
* Subjects may receive other systemic anti-tumor therapies during the study period.
* known allergy to Fluzoparib, apatinib and its excipients.
* In the investigator's judgment, the subjects have other factors that may lead to the forced termination of the study, such as other serious medical conditions (including mental illness) requiring combined treatment, serious laboratory abnormalities, family or social factors that may affect the safety of the subjects, or the collection of data and samples.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival(PFS) | Up to 2 years
  To determine the efficacy by progression free survival (PFS) of the maintenance treatment in previous PARP inhibitor treated platinum-sensitive relapsed ovarian cancer patients according to RECIST v1.1 criteria (Investigator determined).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
Disease Control Rate (DCR） | Up to 2 years
Overall survival (OS） | Up to 2 years
Adverse Events (AEs) | From the first drug administration to within 30 days for the last treatment dose
  Assese the safety and tolerability of Fluzoparib combined with apatinib maintenance in platinum sensitive relapsed ovarian cancer patients by record the number of participants with of AEs and SAEs, and the proportion of patients with AEs and SAEs, etc.

IPD SHARING:
Plan to Share IPD: No
Data is available per require after approved by ethics broad